CLINICAL TRIAL: NCT01909921
Title: Retrospective Medical Record Review of Mind Body Depression Group Participants
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, John W. Denninger, MD, PhD, Director of Research at the Benson-Henry Institute for Mind Body Medicine, Massachusetts General Hospital
Other Study IDs: 2010P001513
Record Dates: First submitted 2013-05-28; First posted 2013-07-29 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the effectiveness of a Relaxation Response Intervention for Depression offered to low income populations at Massachusetts General Hospital (MGH) - Chelsea, Revere and Charlestown health centers.

DETAILED DESCRIPTION:
This is a retrospective review of medical records. The study aims to evaluate the effects of participation in the Relaxation Response Intervention for Depression Clinical groups, on patient measures of: 1) depression, anxiety and perceived stress; 2) work productivity and activity impairment; 3) demand for, and adherence to behavioral medicine; 4) medication use for depression and/or anxiety; and 5) dose-response effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving care through MGH-Health Centers
* a diagnosis of depression and/or anxiety
* 21 years of age or older

Exclusion Criteria:

-

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MGH-Health Center patients who have participated in the Relaxation Response Intervention for Depression groups.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Depression scales (CES-D 10) at 8 weeks | Pre- and Post-Intervention (8 weeks)
Change from baseline Anxiety Scales (STAI-20) at 8 weeks | Pre- and Post- Intervention (8 weeks)
Change from baseline in Perceived Stress Scale (PSS-10) at 8 weeks | Pre- and Post-Intervention (8 weeks)